CLINICAL TRIAL: NCT06380075
Title: COmparison of Clarus and Optos Ultrawide Field Imaging Systems for Inherited Retinal Disease
Acronym: COCO-IRD
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Wisconsin, Madison (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: 2024-0480; A536000 (Other: UW Madison); SMPH/OPHTHAL&VIS SCI/GEN (Other: UW Madison); Protocol Version 3/22/24 (Other: UW Madison)
Record Dates: First submitted 2024-04-18; First posted 2024-04-23 (Actual); Last update posted 2025-12-26 (Actual); Status verified 2025-04

CONDITIONS: Retinal Disease
MeSH Terms: conditions — Retinal Diseases

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

ARMS (1):
- Fundus autofluorescence (FAF) imaging (Experimental)
  Interventions: Device: Spectralis FAF imaging; Device: Optos imaging; Device: Clarus imaging

INTERVENTIONS:
Device: Spectralis FAF imaging — Spectralis is a scanning laser ophthalmoscope which uses a blue light excitation wavelength of 488nm and a 500nm barrier filter to produce FAF images. Spectralis images 20-55 degrees of the retina.
Device: Optos imaging — Optos is an ultrawide field imaging platform which images up to 200 degrees of the retina. It uses both a green-light excitation wavelength of 532nm and a red-light excitation wavelength of 633nm with an emission filter of greater than 540nm to produce FAF images.
Device: Clarus imaging — Clarus 700 is an ultrawide field imaging system with similar retinal coverage to that of Optos. It uses Broad Line Fundus Imaging to produce blue FAF images at excitation wavelengths of 435-500nm and green FAF images at wavelengths of 500-585nm

SUMMARY:
The goal of this research study is to compare two ultrawide field cameras to the gold standard imaging system to evaluate the back of the eye. The main question it aims to answer is the same results and information can be acquired from all of the cameras for evaluating and monitoring inherited retinal diseases (IRDs).

Participants will:

* undergo pupillary dilation
* have photographs taken of the inside of the eyes using three different cameras

ELIGIBILITY:
Inclusion Criteria:

* Participants 18 years and older with a clinical and/ or genetic diagnosis of IRD recruited either from the clinic and/or the Inherited Ocular Disease Registry to participate in this trial
* Participants that are willing to participate as evidenced by signing the written informed consent

Exclusion Criteria:

* Presence of ocular conditions other than an IRD which may affect the quality of ocular imaging including but not limited to advanced cataracts, corneal disorders, nystagmus, vitreous hemorrhage, or poor dilation
* Presence of ocular conditions other than an IRD which may affect interpretation of retinal imagining including but not limited to epiretinal membrane, choroidal neovascular membrane, or macular scarring
* Patients with advanced IRDs who are unable to fixate for imaging
* Patients unable to tolerate ocular imaging
* Patients who do not wish to participate

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Estimated)
Dates: Start 2024-08-29 (Actual); Primary Completion 2026-12 (Estimated); Study Completion 2026-12 (Estimated)

PRIMARY OUTCOMES:
Compare FAF retinal patterns by Clarus and standard Spectralis FAF imaging | Up to 2 hours
  Graders will independently measure area of FAF retinal patterns from images of each device. The measurements (in mm²) will be compared between the two devices.
Compare FAF retinal patterns by Optos and standard Spectralis FAF imaging | Up to 2 hours
  Graders will independently measure area of FAF retinal patterns from images of each device. The measurements (in mm²) will be compared between the two devices.
Compare FAF retinal patterns by Clarus and Optos FAF imaging | Up to 2 hours
  Graders will independently measure area of FAF retinal patterns from images of each device. The measurements (in mm²) will be compared between the two devices.
Compare Spectralis FAF imaging to Spectralis OCT imaging | Up to 2 hours
  In participants with clearly defined macular FAF retinal pattern changes, graders will independently measure area of retinal patterns from images of each device. The measurements (in mm²) will be compared between the two devices.

SECONDARY OUTCOMES:
Prevalence of FAF retinal pattern changes beyond the standard 30 degress in Clarus and Optos ultrawide field images | Up to 2 hours
  The presence of FAF retinal pattern changes outside field 2 will be documented from the two ultrawide field imaging devices
Prevalence of other autofluorescence abnormalities unique to the IRD across all imaging | Up to 2 hours
  The presence of abnormal autofluorescence outside field 2 will be documented from the two ultrawide field imaging devices

CONTACTS AND LOCATIONS:
Overall Officials: Kimberly Stepien, MD, Principal Investigator — University of Wisconsin, Madison
Locations (1):
- Department of Ophthalmology and Visual Sciences, Madison, Wisconsin, United States

IPD SHARING:
Plan to Share IPD: No